CLINICAL TRIAL: NCT01303250
Title: Balanced 6 % HES 130/0.4 vs. Balanced Crystalloid-based Infusion in Patients Undergoing Colorectal Surgery
Brief Title: Perioperative Colloid vs Crystalloid in Patients Undergoing Colorectal Surgery
Acronym: KoKris
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The final decision of the review of HES-containing solution shall be awaited.
Sponsor: University Hospital Muenster (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKM09_0031; 2009-017595-25 (EudraCT Number); 04-AnIt-09 (Other: Department of Anesthesiology, University Hospital Muenster)
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Surgery, Colorectal
Keywords: goal-directed fluid optimization; hemodynamic optimization; crystalloid; colloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): A balanced hydroxyethyl starch 130/0.4 will be used
  Interventions: Drug: balanced 6% hydroxyethylstarch 130/0.4
- Group 2 (Active Comparator): A balanced crystalloid will be used
  Interventions: Drug: balanced crystalloid

INTERVENTIONS:
Drug: balanced 6% hydroxyethylstarch 130/0.4 — Fluid administration and optimization based on cardiac output findings during surgery.
  Arms: Group 1
Drug: balanced crystalloid — Fluid administration and optimization based on cardiac output findings during surgery.
  Arms: Group 2

SUMMARY:
The primary purpose of this study is to determine the effect of a balanced 6%hydroxyethyl starch 130/0.4 vs. a balanced crystalloid in colorectal surgery. The intraoperative fluid management will be given to optimize the stroke volume variation <= 12%.

The investigators hypothesize that patients in the intervention group will need less fluid administration be optimal hemodynamic stabilized.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective colorectal surgery
* minimum age 18 years
* informed consent

Exclusion Criteria:

* patients with severe cardiomyopathy or severe heart failure
* history of coagulation disorders
* intracranial hemorrhage
* patients with severe cardiovascular or respiratory disorders
* renal insufficiency
* severe liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Total amount of administered fluids | intraoperatively
  Total amount of administered fluids intraoperatively that is necessary to keep patients optimal hemodynamic stabilized

SECONDARY OUTCOMES:
Incidence of surgery related complications | day 28 and 90 postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Van Aken, Prof. MD, Principal Investigator — Department of Anesthesia and Intensive Care, University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany